CLINICAL TRIAL: NCT06890130
Title: Long-Term Outcomes of Fracture Odontoid Management in Assiut University
Brief Title: Outcomes of Fracture Odontoid Management
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdelwahab Hassan Hasanien, resident Orthopaedic and Trauma Surgery, Assiut University
Other Study IDs: Outcomes Of Fracture Odontoid
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Odontoid Fracture
Keywords: odontoid fracture; management; long term outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All patients with odontoid fractures presenting to Assiut University Hospital - Department of Orthop: This population likely includes individuals of various ages and backgrounds who have experienced trauma leading to this specific type of fracture. The study may focus on patients who have undergone different treatment strategies, such as surgical intervention or conservative management, to assess the effectiveness and outcomes of these approaches over time. The demographic characteristics of the population could include age, gender, cause of injury, and pre-existing health conditions, which might influence treatment outcomes.

SUMMARY:
This study aims to evaluate the long-term outcomes of treating patients with odontoid fractures admitted to the Trauma Unit of Assiut University Hospital.

DETAILED DESCRIPTION:
study focuses on assessing the long-term results of treatment for patients diagnosed with odontoid fractures. These fractures involve the odontoid process of the second cervical vertebra and can be serious due to their potential impact on spinal stability and neurological function. The study is conducted within the Trauma Unit of Assiut University Hospital, indicating that it involves patients who have been admitted for acute care following such injuries. The long-term outcomes likely include factors such as recovery rates, complications, and the effectiveness of different treatment modalities.

The study population consists of patients admitted to the Trauma Unit of Assiut University Hospital with diagnosed odontoid fractures. This population likely includes individuals of various ages and backgrounds who have experienced trauma leading to this specific type of fracture. The study may focus on patients who have undergone different treatment strategies, such as surgical intervention or conservative management, to assess the effectiveness and outcomes of these approaches over time. The demographic characteristics of the population could include age, gender, cause of injury, and pre-existing health conditions, which might influence treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All patients with odontoid fractures presenting to Assiut University Hospital - Department of Orthopaedic and Trauma Surgery who have completed a minimum of 2 year follow up regardless of age, mechanism of injury, neurological status or type of treatment applied.

Exclusion Criteria:

* • Patients who are not available for two year follow-up

  * Patients who refuse to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients admitted to the Trauma Unit of Assiut University Hospital with diagnosed odontoid fractures. This population likely includes individuals of various ages and backgrounds who have experienced trauma leading to this specific type of fracture. The study may focus on patients who have undergone different treatment strategies, such as surgical intervention or conservative management, to assess the effectiveness and outcomes of these approaches over time. The demographic characteristics of the population could include age, gender, cause of injury, and pre-existing health conditions, which might influence treatment outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of improvement | 2 years
  Percentage of improvement in NDI following conservative and surgical treatment during the follow up visits

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cutler HS, Guzman JZ, Lee NJ, Kothari P, Kim JS, Shin JI, Leven DM, Cho SK. Short-Term Complications of Anterior Fixation of Odontoid Fractures. Global Spine J. 2018 Feb;8(1):47-56. doi: 10.1177/2192568217698132. Epub 2017 May 16. PMID 29456915